CLINICAL TRIAL: NCT02201199
Title: A Single-Center, Randomized, Double-Blind, 3-Treatment, 3-Period, 6-Sequence Cross-Over Study To Compare The Pharmacokinetic And Pharmacodynamic Effects of Single Doses of Insulin Glargine Given As U200 And U500 To Lantus® In A Euglycemic Clamp Setting In Subjects With Type 1 Diabetes
Brief Title: Single Dose Clamp Study To Compare Concentration/Time Profile And Metabolic Activity Profile Of 2 New Formulations Of Insulin Glargine With Lantus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PDY13928; 2014-001252-33; U1111-1153-3712 (Other: UTN)
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- insulin glargine U100 (Active Comparator): 1 single dose
  Interventions: Drug: insulin glargine U100 HOE901
- insulin glargine U200 (Experimental): 1 single dose
  Interventions: Drug: insulin glargine U200 HOE901
- insulin glargine U500 (Experimental): 1 single dose
  Interventions: Drug: insulin glargine U500 HOE901

INTERVENTIONS:
Drug: insulin glargine U200 HOE901 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Arms: insulin glargine U200
Drug: insulin glargine U500 HOE901 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Arms: insulin glargine U500
Drug: insulin glargine U100 HOE901 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Other Names: Lantus
  Arms: insulin glargine U100

SUMMARY:
Primary Objective:

To compare the pharmacokinetic (PK) characteristics of single doses of insulin glargine given as U200 and U500 with those of a single dose (SD) of Lantus® U100 in a euglycemic clamp setting in subjects with type 1 diabetes.

Secondary Objectives:

To compare the metabolic activity characteristics of single doses of insulin glargine given as U200 and U500 with those of a single dose of Lantus® U100 in a euglycemic clamp setting in subjects with type 1 diabetes.

To assess the safety and tolerability of single doses of U200, U500 and Lantus® U100 in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
Total study duration for each subject is between 3.5 and 12 weeks.

Two overnight stays at the unit in each of 3 treatment periods.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects, between 18 and 65 years of age, inclusive, with type 1 diabetes mellitus for more than one year, as defined by the American Diabetes Association.
* Total insulin dose <1.2 U/kg/day.
* Minimum usual basal insulin dose ≥0.2 U/kg/day.
* Body weight between 50.0 kg and 110.0 kg, Body Mass Index between 18.5 and 30.0 kg/m2 inclusive.
* Fasting negative serum C-peptide (<0.3 nmol/L).
* Glycohemoglobin (HbA1c) ≤75 mmol/mol (≤9.0%).
* Stable insulin regimen for at least 2 months prior to inclusion in study.
* Certified as otherwise healthy for Type 1 diabetes mellitus patient.
* Women of childbearing potential with negative pregnancy test and use of a highly effective contraceptive method or women with confirmed postmenopausal status.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion criteria:

* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months.
* Frequent severe headaches and / or migraine, recurrent nausea and / or vomiting (more than twice a month).
* Presence or history of a drug allergy or clinically significant allergic disease according to the Investigator's judgment.
* Presence or history of drug or alcohol abuse (alcohol consumption >40 grams / day).
* Smoking more than 5 cigarettes or equivalent per day, unable to refrain from smoking.
* Any medication (including St John's Wort) within 14 days before inclusion, or within 5 times the elimination half-life or pharmacodynamic half-life of that drug, whichever the longest and regular use of any medication in the last month before study start with the exception of insulin products, thyroid hormones, lipid-lowering and antihypertensive drugs, and, if female, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days; any biologics (antibody or its derivatives) given within 4 months before randomization.
* Known hypersensitivity to insulin glargine or excipients of the study drug.
* Any history or presence of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in first degree relatives (parents, siblings or children).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin glargine (INS) concentration curve over the first 12 hours after dosing | 12 hours

SECONDARY OUTCOMES:
INS-Area Under the Curve (AUC) over 24 and 36 hours after dosing (INS AUC 0-24 and INS AUC 0-36) | 36 hours
AUC up to the last measurable concentration | 36 hours
Time to reach 50% of INS-AUC 0-36 | 36 hours
Time to reach INS-Cmax (INS-tmax) | 36 hours
Area under the body-weight-standardized Glucose Infusion Rate (GIR) over the first 12, 24 and 36 hours after dosing (GIR-AUC0-12, GIR-AUC0-24 and, GIR-AUC0-36) | 36 hours
Time to reach 50% of GIR-AUC0-36 (T50%-GIR-AUC0-36) | 36 hours
Maximum smoothed body weight standardized glucose infusion rate (GIRmax) and time to GIRmax (GIR-Tmax) | 36 hours
Duration of blood glucose control (time to elevation of smoothed blood glucose profile above different pre-specific blood glucose levels) | 4 days
Safety and tolerability (Number of patients with adverse events, clinically significant changes in vital signs, laboratory parameters) | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Neuss, Germany